CLINICAL TRIAL: NCT05780866
Title: Remote Monitoring in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacob E. Simmering (Other)
Responsible Party: Sponsor-Investigator, Jacob E. Simmering, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202111199
Record Dates: First submitted 2023-03-10; First posted 2023-03-23 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Videotape Recording; Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Video and Activity Tracker (Other)
  Interventions: Other: Video and Activity Tracker

INTERVENTIONS:
Other: Video and Activity Tracker — At enrollment, the participants will complete a baseline survey, PDQ-39 (Parkinson's disease questionnaire), and the Unified Parkinson's Disease Rating Scale (UPDRS) assessment. The researchers will provide the participant with a camera, small tripod, and a set of written directions about how to record the UPDRS motor self-assessment video.
  After completing the baseline assessments, the research team will provide the participant with a Fitbit Inspire 3 activity tracker watch. The participant will wear the activity tracker for 24 hours a day for the next 14 days except for if the device needs charging and when bathing.
  At 14 days, the research team will send participants a link to complete a web-based exit survey about their experience with the activity tracker during the study.

SUMMARY:
The goal of this observational study is to learn about the usefulness of physical activity measures and tremor detection using wearable devices and smartphone video to detect and evaluate disease burden in people with Parkinson's disease.

Participants will wear an activity tracker at home and complete a short research visit where they will make a video using a smartphone of themselves performing a fine motor task. They will wear the activity tracker for two weeks at home.

DETAILED DESCRIPTION:
For all groups (there is no control group):

At enrollment, the participants will complete a baseline survey that records participant sex, years since the diagnosis of Parkinson's disease, current use of levodopa medication, and whether levodopa was taken today.

Next, a research nurse from neurology will complete the Unified Parkinson's Disease Rating Scale (UPDRS) assessment. As part of this assessment, the researchers will make a video recording of Part 3 (the motor assessment) as a gold standard for comparison with the participant-recorded videos.

Next, the participant will complete the PDQ-39 (Parkinson's disease questionnaire), a 39 item questionnaire about the quality of life.

After completing the PDQ-39, the researchers will provide the participant with a camera, small tripod, and a set of written directions about how to perform the UPDRS motor assessment. The goal with this task is to simulate a home recording session to uncover any issues and create preliminary data for validation of the home recording compared to the gold standard collected by the study team. The recordings will then be converted to x, y, z landmarks using MediaPipe, running on UIowa hardware.

After completing the video, the participant will complete a short survey about ease of making the video recording.

After completing the baseline assessments, the research team will provide the participant with a Fitbit Inspire 3 activity tracker watch, configure the tracker to sync with their phone, and provide an overview of use.

The participant will wear the activity tracker for 24 hours a day for the next 14 days except for if the device needs charging and when bathing.

At 14 days, the research team will send participants a link to complete a web-based exit survey about their experience with the activity tracker during the study.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of PD
* Current patient at UIHC Movement Disorders clinic
* Owns a smartphone that is compatible with a activity tracker.

Exclusion Criteria

* Non-English speaking
* Bedridden or uses a wheelchair the majority of the time
* Prisoner status
* Inability to provide own informed consent

Ages: 50 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Activity tracker wear rate | 14 Days
  Percent of time activity tracker records a heart rate
Accuracy of computer vision assessment of motor function | Baseline
  Average difference in UPDRS score between human and computer assessments
Do step counts predict quality-of-life | 14 Days
  Regression of PDQ-39 on demographics and activity tracker step counts

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Simmering, MS, PHD, BA, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States